CLINICAL TRIAL: NCT05995535
Title: Pregabalin Plus Lofexidine for the Outpatient Treatment of Opioid Withdrawal
Acronym: UH3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kyle Kampman, Professor, Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 854046
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Opiate Withdrawal Syndrome; Opioid Use
MeSH Terms: interventions — lofexidine; Pregabalin

STUDY DESIGN:
Intervention Model Description: Active pregabalin plus lofexidine versus placebo pregabalin plus lofexidine
Who Masked: Participant, Investigator
Masking Description: double-blind placebo-controlled randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LFX/PGB (Experimental): PGB/day 1=400mg, day 2-7=600mg each day, day 8=400mg, day 9=200mg, day 10=100mg
  LFX/day 1=1.62mg, day 2-7=2.16mg each day, day 8=1.44mg, day 9=0.72mg, day 10=0.72mg
  Interventions: Drug: LFX/PGB; Drug: LFX/PLA-PGB
- LFX/PLA-PGB (Active Comparator): PLA-PGB/day 1-7= 0mg each day, day 8, 9, and 10 =0mg each day
  LFX/ day 1=1.62mg, day 2-7=2.16mg each day, day 8=1.44mg, day 9=0.72mg, day 10=0.72mg
  Interventions: Drug: LFX/PGB; Drug: LFX/PLA-PGB

INTERVENTIONS:
Drug: LFX/PGB — lofexidine tablets 0.18mg tabs
  pregabalin capsules 100mg and 25mg
  Other Names: Lucemyra; lyrica
Drug: LFX/PLA-PGB — lofexidine tablets 0.18mg tabs
  pregabalin capsules 0mg
  Other Names: Lucemyra; placebo pregabalin

SUMMARY:
A placebo-controlled trial in which male and female outpatients with an opioid use disorder who express interest in extended-release injectable naltrexone (XR-NTX) are randomized 1:1 to lofexidine/pregabalin or lofexidine/pregabalin placebo for withdrawal management and offered XR-NTX if after completing withdrawal.

DETAILED DESCRIPTION:
A placebo-controlled trial in which male and female outpatients with an opioid use disorder who express interest in extended-release injectable naltrexone (XR-NTX) are randomized 1:1 to lofexidine/pregabalin or lofexidine/pregabalin placebo for withdrawal management and offered XR-NTX if after completing withdrawal. It follows a UG3 study in which 90 inpatients with an OUD who expressed interest in XR-NTX were randomized 2:1 to withdrawal management with lofexidine/pregabalin or lofexidine/placebo pregabalin. Results were that the conditions were equally safe, and that lofexidine/pregabalin was more effective in reducing subjective withdrawal and keeping patients in treatment than lofexidine/placebo pregabalin.

The objectives are to study the safety and effectiveness of lofexidine/pregabalin compared to lofexidine/placebo for managing opioid withdrawal and transitioning to XR-NTX in outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects ≥ 18 years of age
2. Meet DSM-5 criteria for an Opioid Use Disorder with physiologic features. Have met 2 or more of the 11 criteria for an OUD including tolerance and withdrawal within the last 12 months
3. Interested in opioid antagonist treatment
4. Used opioids in 20 or more of the last 30 days
5. A stable address in the local area; not planning to move in the next 60 days.
6. Have documents for ID check
7. Absence of medical or psychiatric conditions that are likely to interfere with study participation
8. Has 12 lead ECG demonstrating a QTc ≤450 msec and a QRS ≤120 msec. Site PI has final determination for study inclusion if readings exceed these limits. The PENN cardiologists and medical monitor are available for consultation when needed
9. Negative pregnancy test and using adequate contraception if of childbearing potential.

Exclusion Criteria:

1. Current psychotic disorder (bipolar I, schizophrenia, major depression that is not in remission
2. Alcohol, benzodiazepine, or other sedative use disorder with physiological features that require medication for detoxification
3. Allergy or other serious adverse event due to treatment with pregabalin, XR-NTX, or lofexidine
4. Pending incarceration or plans to leave the immediate area in the next 30 days
5. Homicidal or otherwise behaviorally disturbed requiring immediate attention
6. High risk for suicide as determined by answering 'yes' to questions 4 and/or 5 on C-SSRS
7. Blood pressure <90 mm Hg (systolic) or <60 mm Hg (diastolic). If value out of normal range, the investigator and study Clinician will decide subject inclusion/exclusion on case-by-case basis
8. Heart rate and/or pulse<50 bpm at screening-sitting
9. An Estimated Glomerular Filtration Rate eGFR<70 mL/min/1.73m2
10. A History of, or current Seizure disorder (excluding childhood febrile seizures)
11. Inability to read and/or understand English. For example, unable to understand the informed consent as demonstrated by failing to answer 9/10 questions correctly on the quiz
12. 12. Pregnant or breastfeeding
13. 13. Currently taking sympathomimetic drugs, or a thiazolidinedione antidiabetic
14. ALT and/or AST >4X upper limit of normal
15. A Child-Pugh score >7
16. Currently receiving opioids for pain management
17. In a treatment study where medication was administered in the last 30 days
18. Currently using medications that are known to be strong or moderate inhibitors of CYP2D6 such as fluoxetine, paroxetine, mirabegron, bupropion, quinidine, terbinafine, cimetidine, cinacalcet, duloxetine, or fluvoxamine
19. In a methadone maintenance or buprenorphine treatment program within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Opioid Withdrawal Scale (SOWS) scores | 10 days per subject, through study completion (N=150)
  Subjective patient reported Opioid Withdrawal measured by the SOWS, (0-30); 0 = no withdrawal/30 = severe withdrawal

SECONDARY OUTCOMES:
Study detox completion | 10 days per subject, through study completion (N=150)
  Proportion that receives one or more doses of study medication and completed withdrawal (Completing withdrawal management will be defined as having received at least 1 dose of study medication on day 8 and completing the SOWS-Gossop assessment on day 8); and proportion that transition to XR-NTX; adverse events
XR-NTX IM injection | upto 2 days per subject (N=150)
  proportion that receives 380mg dose of extended-release naltrexone

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mountain Manor Treatment Center, Baltimore, Maryland
  - University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No